CLINICAL TRIAL: NCT01924884
Title: Surgical Site Infection (SSI) Rate After Intra-Abdominal Surgery Using Negative Pressure Wound Therapy (NPWT) at Initial Closure
Brief Title: Surgical Site Infection Rate After Intra-Abdominal Surgery Using Negative Pressure Wound Therapy at Initial Closure
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Kinetic Concepts, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB00155110; NA_00052186 (Other: Other)
Record Dates: First submitted 2013-08-05; First posted 2013-08-19 (Estimated); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Surgical Wound Infection; Wound; Abdomen, Abdominal Wall; Surgery
Keywords: Vacuum-Assisted Closure; Topical Negative-Pressure Therapy; Negative-Pressure Dressings
MeSH Terms: conditions — Surgical Wound Infection; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Prospective: Patients newly referred to the Principal Investigator for intra-abdominal surgery and for whom the Principal Investigator anticipates using Negative-Pressure Wound Therapy.
- Retrospective: Patients who underwent intra-abdominal surgery by the Principal Investigator between January 1, 2011 and May 9, 2013 will be identified through patient medical records. Living patients will be contacted via letter from the Principal Investigator introducing the study along with the study's consent form for the patients' review. Interested patients will be consented either in person at the patient's next clinic visit or via telephone by a member of the study staff.
- Historical Controls: Patients who underwent intra-abdominal surgery without Negative-Pressure Wound Therapy by the Principal Investigator prior to January 1, 2011 will be enrolled as Historical Controls.
- De-Identified Retrospective: Patients who underwent intra-abdominal surgery by the Principal Investigator between January 1, 2011 and May 9, 2013 and are deceased or do not consent to be in the study will be enrolled in the De-Identified Retrospective Case Cohort.

SUMMARY:
The goal of this study is to present a large single-institution experience reporting surgical site infection rates in patients who have undergone intra-abdominal surgery followed by wound closure with Negative Pressure Wound Therapy. A retrospective review of patients' charts will be conducted to analyze surgical site infection rates between wound closure with and without Negative Pressure Wound Therapy (NPWT). American College of Surgeons National Quality Improvement Program data from previous standard of care (primary closure after colorectal surgery) will be used for comparison with newly adopted standard of care treatment regimen (wound closure with NPWT).

Data on patients who underwent intra-abdominal surgery will be retrospectively collected and a database will be created. These individuals will be identified through medical records and recontacted by mail and/or phone to collect study data.

Finally, patients newly referred to the Principal Investigator for intra-abdominal surgery will be enrolled in the database. After giving informed consent, data on surgical site infection rates and outcomes will be collected. Longitudinal outcomes will be assessed at 30 days, 6 months, and 12 months post-operatively. These patients' outcomes will be compared to a group of patients treated by the Principal Investigator who also underwent intra-abdominal surgery without Negative Pressure Wound Therapy. We hypothesize that fewer patients treated with negative pressure wound therapy following intra-abdominal surgery will develop surgical site infections than patients who had intra-abdominal surgery but were not treated with Negative Pressure Wound Therapy.

DETAILED DESCRIPTION:
Duration of individual study participation will last approximately one year for prospectively enrolled participants. Data collection for retrospectively enrolled patients will span approximately 12 months.

Study data will not be collected on subjects until eligibility is confirmed and the patient is assigned a study number.

All information will be collected in a secure study-specific electronic registry database. The data will be reviewed for completeness and accuracy by the Principal Investigator. This is an observational registry which does not include an investigatory agent and poses minimal risk to the participants. Thus, the monitoring will be done by the study personnel - an independent board is not necessary.

This study will use the descriptions and grading scales found in the revised National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 4. Information about all adverse events, whether volunteered by the subject, discovered by the investigator, or detected through physical examination, laboratory test, or other means, will be collected, recorded, and followed as appropriate. All adverse events experienced by participants will be collected and reported from the time of consent until the Day 30 follow-up appointment, as appropriate. Thereafter, only adverse events of interest (i.e., death, additional hospitalization, surgical site infection, surgical site occurrence) will be recorded. Participants who have an ongoing adverse event related to the study procedures may continue to be periodically contacted by a member of the study staff until the event has resolved or determine to be irreversible by the principal investigator. All adverse events and serious adverse events will be reported to the Johns Hopkins Medicine Institutional Review Board.

To generate a large data set that may be used to answer various research questions, enrollment will continue for at least 10 years, generating an estimated patient sample size of n=1200. The study team anticipates enrolling 100-150 patients in the study registry per year over 10 years.

Simple descriptive statistics will be used to determine the rate of SSIs in colorectal surgery patients. This rate will be compared with the SSI rate published in literature to determine if implementation of negative pressure wound therapy wound closure following colorectal surgery decreases the rate of SSIs in colorectal surgery patients. A hypothesis test will be used to determine if there is a difference before and after adoption of negative pressure wound therapy wound closure. Enrollment of subjects over several years will enable further analyses with the possibility of stratification according to different patient characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years of age
* Undergoing intra-abdominal surgery at Johns Hopkins Hospital by Dr. Frederic Eckhauser

Exclusion Criteria:

* Less than 18 years of age
* Pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients greater than or equal to 18 years of age undergoing intra-abdominal surgery at Johns Hopkins Hospital by Dr. Frederic Eckhauser. Both men and women and members of all races and ethnic groups are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Surgical site infection (per the 1999 Guideline for Prevention of Surgical Site Infection from the Hospital Infections Program at the National Center for Infectious Diseases, Centers for Disease Control and Prevention). | Up to one year
  Comparing surgical site infection (per the 1999 Guideline for Prevention of Surgical Site Infection from the Hospital Infections Program at the National Center for Infectious Diseases) rates between patients treated with and without negative pressure wound therapy.
  Objective: To determine if a newly adopted standard of care [negative pressure wound therapy (NPWT)] for clean, clean-contaminated, and contaminated wounds will lead to decreased rates of post-operative surgical site infection.

SECONDARY OUTCOMES:
Surgical site occurrence (per the 2010 Ventral Hernia Working Group's classification and the modified hernia grading scale by Kanters et al.; 2012). | Up to one year
  Comparing surgical site occurrence (per the 2010 Ventral Hernia Working Group's classification and the modified hernia grading scale by Kanters et al.; 2012) rates between patients treated with and without negative pressure wound therapy.
  Objective: To determine if a newly adopted standard of care [negative pressure wound therapy (NPWT)] for clean, clean-contaminated, and contaminated wounds will lead to decreased rates of post-operative surgical site occurrence.
Quantifying post-operative morbidity and mortality rates among patients undergoing bowel surgery with or without negative pressure wound therapy. | Up to one year
  Objective: To determine if a newly adopted standard of care [negative pressure wound therapy (NPWT)] for clean, clean-contaminated, and contaminated wounds will improve outcomes of bowel surgery patients.

OTHER OUTCOMES:
Quantifying post-operative morbidity and mortality rates among patients undergoing enterocutaneous fistula and ventral hernia repair with or without negative pressure wound therapy. | Up to one year
  Objective: To determine morbidity and mortality secondary to enterocutaneous fistula and ventral hernia repair in this patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Carisa Cooney, MPH, CCRP, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Pooled data will be shared.